CLINICAL TRIAL: NCT06723262
Title: Contribution to Speech Perception of a Tonotopy-based Fitting for Patients With Cochlear Implants for 6 Months With a Conventional Setting: Prospective Cross-sectional Study
Brief Title: Speech Perception of a Tonotopy-based Fitting for Cochlear Implant Recipients for 6 Months With Conventional Setting
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MED-EL Elektromedizinische Geräte GesmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MEDEL_ABF6m_Limoges_study
Record Dates: First submitted 2024-12-04; First posted 2024-12-09 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Sensorineural Hearing Loss, Bilateral
Keywords: cochlear implant strategy anatomy-based fitting
MeSH Terms: conditions — Hearing Loss, Sensorineural

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ABF arm (Other): At 6 month post-activation: tonotopic fitting FS4T the participant wears FS4T during 6 weeks.
  Interventions: Other: Tonotopic cochlear implant fitting FS4T

INTERVENTIONS:
Other: Tonotopic cochlear implant fitting FS4T — Comparison of FS4T and FS4noT
  Other Names: No tonotopic cochlear implant fitting FS4noT

SUMMARY:
Main objective:

Compare speech recognition in noise with tonotopic fitting (FS4T) and with conventional non-tonotopic fitting (FS4noT) in adult patients implanted for 6 months with a MED-EL cochlear implant with FS4noT strategy.

Secondary objectives:

Comparison of FS4noT and FS4T settings

* for speech recognition in quiet
* for subjective auditory spatial perception

DETAILED DESCRIPTION:
Introduction: Cochlear implantation allows the rehabilitation of profound bilateral deafness, restoring speech perception and verbal communication when the traditional hearing aid no longer provides satisfactory hearing gain. A cochlear implant includes an electrode array and its functioning is based on the principle of cochlear tonotopy: each electrode encodes a frequency spectrum according to its position in the cochlea (high frequencies are assigned to the basal electrodes and low frequencies to the apical electrodes). The cochlear implant thus breaks down the frequency spectrum into a number of frequency bands via bandpass filters corresponding to the number of electrodes in the implant. During the fitting these bands can be modified by the audiologist. The fitting software developed by the manufacturers proposed a default fitting with a lower limit between 100 and 250 Hz according to the brands and an upper limit of about 8500 Hz. The frequency bands assigned to each electrode follow a logarithmic scale with the high frequencies for the basal electrodes and the low frequencies for the apical electrodes. This distribution takes into account the number of active electrodes but does not take into account the anatomy and the natural cochlear tonotopy specific to each patient. Several studies have analyzed the anatomical variations of the cochlear dimensions: size of the cochlea and the ratio between the contact surfaces of the electrodes with the cochlea are variable from one patient to another. The insertion depth during surgery is also variable due to parameters related to the patients as well as to the operator, which seems to impact the understanding of speech in noise. Mathematical algorithms have recently been developed to estimate the cochlear tonotopy of each patient from a CT scan assessment. CT imaging of the implanted ear combined with 3D reconstruction software, provides cochlear length measurements. Using this approach it is possible to measure the position of each electrode relative to the cochlear apex. Recently, MED-EL (Austria) has developed a new approach based on CT-scan and tuning of the frequencies associated with each electrode using anatomical information of position of the electrodes in the cochlea: this fitting is called anatomy-based fitting (ABF).

Recently [Jiam et al. 2016, 2019] showed that a frequency fitting based on the tonotopy of the electrodes allowed to obtain a better perception of pitch after 30 minutes of acclimatization. In a prospective randomized crossover study with a wearing time of 6 weeks on new cochlear implantees, Creff et al. (2023, 2024) obtained very significantly superior results with a tonotopic setting compared to a classic setting (HDCIS) for speech recognition tests in noise and for musical perception. However, even if the tonotopic setting appears particularly promising over a period of 6 weeks, it is possible that the difference diminishes over time (Mertens et al.,2021). Brain plasticity could partially or completely compensate for the mismatch after a few months/years of CI use (Svirsky et al. 2004; Reiss et al. 2007, 2014). However, this adaptation may remain incomplete or prolong the acclimatization period even after numerous rehabilitation sessions (Sagi et al. 2010; Svirsky et al. 2015; Tan et al. 2017; Dorman et al. 2022). Further studies on the use of tonotopy-based fitting and its effects on speech understanding, also in experienced CI users, are therefore needed.

Main objective:

Compare speech recognition in noise with tonotopic fitting (FS4T) and with conventional non-tonotopic fitting (FS4noT) in adult patients implanted for 6 months with a MED-EL cochlear implant with FS4noT strategy.

Secondary objectives:

Comparison of FS4noT and FS4T settings

* for speech recognition in quiet
* for subjective auditory spatial perception

Plan of the study: It is a prospective open monocentric transversal study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (>= 18 years old) speaking French
* Patient who fulfils the criteria for cochlear implantation

Exclusion Criteria:

* retro-cochlear pathology: auditory neuropathy, vestibular schwannoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Speech recognition in noise | 6 weeks after FS4T fitting
  Framatrix test. Speech and noise in front the participant (at 1m). Noise level: 65 dB SPL. Speech level: adaptive with the answers of the participant. Result: speech-to-noise ratio (speech reception threshold, SRT50) for 50% of intelligibility in noise.
  Test with FS4T and with FS4noT

SECONDARY OUTCOMES:
Speech recognition in quiet | 6 weeks after FS4T fitting
  Two lists of 10 disyllabic words (Fournier lists) at 65 dB SPL. The participant has to repeat the word emitted. Result: score on 20.
  Test with FS4T and with FS4noT.
Subjective auditory spatial perception | At FS4T fitting and 6 weeks after FS4T fitting
  Questionnaire SSQi15 (" Speech, Spatial, and Qualities of hearing scale ", SSQ). The questionnaire consists of 15 questions describing various real-world hearing situations.
  The subject answers each question with a score on a visual analogue scale graduated from 0 (worse) to 10 (better) ranging from "not at all" (0) to "yes perfectly" (10).
  The result obtained is composed of
  * a total average score equal to the sum of the scores of all the questions divided by the total number of questions.
  * 3 average sub-scores describing 3 subscales: Speech hearing with 5 questions Spatial hearing with 5 questions Quality of hearing with 5 questions. Questionnaire with FS4T (at FS4T fitting) and with FS4noT (6 weeks after FS4T fitting)

CONTACTS AND LOCATIONS:
Overall Officials: Karine Aubry, Pr, Principal Investigator — University Hospital, Limoges
Locations (1):
- CHU, Limoges, France

IPD SHARING:
Plan to Share IPD: No